CLINICAL TRIAL: NCT03835143
Title: the Effect of Sub-inguinal Varicocelectomy in Patients Complaining of Orchialgia With Normal Semen Analysis
Brief Title: Outcome of Sub-inguinal Varicocelectomy on Normal Semen in Patients Complaining of Orchilagia With Normal Semen
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdelkader, resident of urology, Assiut University
Other Study IDs: varicocle pain
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Varices; Cord
MeSH Terms: conditions — Varicose Veins; Cone-Rod Dystrophies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: subinguinal varicocelectomy — varicocele ligation done at the level of subinguinal region

SUMMARY:
varicoclelectomy is done for subfertiltiy and varicocele induced orchialgia. The effect of varicocelectomy on semen analysis is controversial. Many articles report favorable outcomes and others do not.

Most study don't focus on varicocelectomy done for varicocele induced orchialgia,and those studies dont report on postoperative semen.

This study will focus on the effect of operation on the semen postoperatively .

ELIGIBILITY:
Inclusion Criteria:

1. Primary varicocele.
2. Patient's age more than 20 years.
3. Scrotal pain (after exclusion of other causes).
4. Normal semen analysis

Exclusion Criteria:

1. Secondary varicocele.
2. Recurrent varicocele.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: there is no description
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Grades of Motility of sperm in semen analysis | 3 months after the operation
  semen analysis

SECONDARY OUTCOMES:
Count of sperms in semen analysis | 3 months after the operation
  semen analysis

OTHER OUTCOMES:
Pain improvement using Numeric Pain Rating Scale | 3 months after the operation
  semen analysis
duppler | 3 months after the operation
  doppler will be done to evaluate the veins pre and postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit Medical School, Asyut, Assuit, Egypt

REFERENCES:
- [Result] Cayan S, Shavakhabov S, Kadioglu A. Treatment of palpable varicocele in infertile men: a meta-analysis to define the best technique. J Androl. 2009 Jan-Feb;30(1):33-40. doi: 10.2164/jandrol.108.005967. Epub 2008 Sep 4. PMID 18772487
- [Result] Kupis L, Dobronski PA, Radziszewski P. Varicocele as a source of male infertility - current treatment techniques. Cent European J Urol. 2015;68(3):365-70. doi: 10.5173/ceju.2015.642. Epub 2015 Oct 15. PMID 26568883
- [Result] Shabana W, Teleb M, Dawod T, Elsayed E, Desoky E, Shahin A, Eladl M, Sorour W. Predictors of improvement in semen parameters after varicocelectomy for male subfertility: A prospective study. Can Urol Assoc J. 2015 Sep-Oct;9(9-10):E579-82. doi: 10.5489/cuaj.2808. Epub 2015 Sep 9. PMID 26425217
- [Result] Paick S, Choi WS. Varicocele and Testicular Pain: A Review. World J Mens Health. 2019 Jan;37(1):4-11. doi: 10.5534/wjmh.170010. Epub 2018 May 16. PMID 29774668
- [Result] Cho CL, Esteves SC, Agarwal A. Novel insights into the pathophysiology of varicocele and its association with reactive oxygen species and sperm DNA fragmentation. Asian J Androl. 2016 Mar-Apr;18(2):186-93. doi: 10.4103/1008-682X.170441. PMID 26732105